CLINICAL TRIAL: NCT03562416
Title: Nintedanib Plus Usual Transplant Care Compared to Usual Transplant Care Alone After Single Lung Transplantation in Patients With Idiopathic Pulmonary Fibrosis: a Pilot Randomized Controlled Trial
Brief Title: Continuation of Nintedanib After Single Lung Transplantation in IPF Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Temple University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1199-0329
Record Dates: First submitted 2018-05-07; First posted 2018-06-19 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Idiopathic Pulmonary Fibrosis; Lung Transplant; Complications
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — nintedanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nintedanib (Experimental): Nintedanib 150 mg tablet by mouth twice daily for 24 months.
  Interventions: Drug: Nintedanib
- Placebo (Placebo Comparator): Placebo tablet by mouth twice daily for 24 months
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Nintedanib — Nintedanib (BIBF 1120, Ofev)
  Other Names: BIBF 1120; Ofev
  Arms: Nintedanib
Drug: Placebo Oral Tablet — Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to assess the utility of nintedanib therapy in addition to usual transplant care in single lung transplant recipients with idiopathic pulmonary fibrosis (IPF). The investigators hypothesize that in IPF subjects who undergo single lung transplantation the administration of nintedanib 150 mg twice daily in addition to usual transplant care will result in better preservation of lung function at 24 months.

DETAILED DESCRIPTION:
Lung transplantation is the only treatment option that augments survival in patients with idiopathic pulmonary fibrosis (IPF). Despite several advancements in lung transplantation over the past three decades, long-term survival rates have remained low compared to other solid organ transplantations. The median survival after lung transplantation is only 5.8 years. Multiple factors account for the relatively low survival post-transplant, but chronic rejection resulting in obliterative bronchiolitis is a predominate cause. Further research is needed to develop medical therapeutic interventions that improve survival in IPF patients who undergo only single lung transplantation.

Nintedanib, a novel tyrosine kinase inhibitor, exhibits antifibrotic properties via multiple mechanisms including the inhibition of the receptor tyrosine kinases platelet derived growth factor (PDGF) receptor, fibroblast growth factor (FGF) receptor, and vascular endothelial growth factor (VEGF) receptor. Several mediators of pulmonary fibrosis including VEGF, FGF, and transforming growth factor beta (TGF-β) have also been implicated in the pathogenesis of bronchiolitis obliterans syndrome (BOS), the most common type of chronic lung allograft rejection.

Nintedanib is safe to continue until the time of lung transplantation and has not been shown to worsen perioperative outcomes in small case series, single center cohorts and our center's personal experience. The current practice in lung transplant medicine is to discontinue antifibrotic therapy after lung transplantation in IPF. In IPF patients who undergo single lung transplant, nintedanib therapy has the potential to preserve lung function in both the native fibrotic lung and the new lung allograft.

The investigators propose a randomized and placebo-controlled single center pilot trial comparing nintedanib therapy plus usual care to usual care only in IPF patients after single lung transplant. The investigators hypothesize that in IPF subjects who undergo single lung transplantation the administration of nintedanib 150 mg twice daily in addition to usual transplant care will result in better preservation of lung function at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 35-70.
* Lung transplantation listing diagnosis of pulmonary fibrosis
* Recipient of single lung transplantation within the past 60 days

Exclusion Criteria:

* History of intolerability to nintedanib (i.e. discontinued nintedanib in the pre-transplant period due to adverse drug effects)
* Liver transaminase elevation (AST or ALT > 1.5X the upper limit of normal)
* Total bilirubin > 1.5X the upper limit of normal
* Drugs that interfere with the metabolism or elimination of nintedanib or its metabolites - St. John's wort, carbamazepine, phenytoin, rifampin, dexamethasone, and others.
* Any history of bronchial anastomosis dehiscence or stenosis
* Bleeding risk, defined as any of the following:

  * Full-dose therapeutic anticoagulation (i.e. vitamin K antagonist, direct thrombin inhibitors, etc.)
  * History of hemorrhagic central nervous system (CNS) event within 12 months of enrollment
  * Coagulation parameters: international normalized ratio (INR) > 2, prolongation of prothrombin time (PT) and partial thromboplastin time (PTT) by > 1.5X the upper limit of normal at enrollment

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Change in FEV1 | Baseline to 24 months
  Change in forced expiratory volume in 1 second (FEV1)
Change in FVC | Baseline to 24 months
  Change in forced vital capacity (FVC)

SECONDARY OUTCOMES:
Bronchiolitis obliterans syndrome | Baseline to 24 months
  Incidence of bronchiolitis obliterans syndrome (BOS)
Bronchial stenosis | Baseline to 24 months
  Incidence of surgical anastomosis bronchial stenosis
Bronchial dehiscence | Baseline to 24 months
  Incidence of surgical anastomosis bronchial stenosis
Acute cellular rejection | Baseline to 24 months
  Incidence of acute cellular rejection of lung allograft
Drug discontinuation | Baseline to 24 months
  Study drug discontinuation rate due to adverse drug event
Adverse drug events | Baseline to 24 months
  Incidence of adverse drug events (i.e. elevation of liver transaminases greater than 3 times the upper limit of normal, diarrhea, nausea, vomiting, anorexia, GERD)
Vascular endothelial growth factor (VEGF) - serum | Baseline to day 30
  Change in serum biomarker concentration for VEGF (pg/mL)
Vascular endothelial growth factor (VEGF) - BAL | Baseline to day 30
  Change in BAL concentration for VEGF (pg/mL)
Vascular endothelial growth factor (VEGF) - serum | Baseline to day 300
  Change in serum concentration for VEGF (pg/mL)
Vascular endothelial growth factor (VEGF) - BAL | Baseline to day 300
  Change in BAL concentration for VEGF (pg/mL)
Fibroblast growth factor (FGF) - serum | Baseline to day 30
  Change in serum concentration for FGF (pg/mL)
Fibroblast growth factor (FGF) - BAL | Baseline to day 30
  Change in BAL concentration for FGF (pg/mL)
Fibroblast growth factor (FGF) - serum | Baseline to day 300
  Change in serum concentration for FGF (pg/mL)
Fibroblast growth factor (FGF) - BAL | Baseline to day 300
  Change in BAL biomarker concentration for FGF (pg/mL)
Platelet derived growth factor (PDGF) - serum | Baseline to day 30
  Change in serum concentration for PDGF (pg/mL)
Platelet derived growth factor (PDGF) - BAL | Baseline to day 30
  Change in BAL biomarker concentration for PDGF (pg/mL)
Platelet derived growth factor (PDGF) - serum | Baseline to day 300
  Change in serum biomarker concentration for PDGF (pg/mL)
Platelet derived growth factor (PDGF) - BAL | Baseline to day 300
  Change in BAL biomarker concentration for PDGF (pg/mL)
Peripheral blood flow cytometry - CD4 T cells | Day 30
  CD4 T cell concentration in peripheral blood (cells/µL)
Peripheral blood flow cytometry - CD4 T cells | Day 300
  CD4 T cell concentration in peripheral blood (cells/µL)
Peripheral blood flow cytometry - CD8 T cells | Day 30
  CD8 T cell concentration in peripheral blood (cells/µL)
Peripheral blood flow cytometry - CD8 T cells | Day 300
  CD8 T cell concentration in peripheral blood (cells/µL)
Peripheral blood flow cytometry - macrophages | Day 30
  Macrophage concentration in peripheral blood (cells/µL)
Peripheral blood flow cytometry - macrophages | Day 300
  Macrophage concentration in peripheral blood (cells/µL)
Peripheral blood flow cytometry - neutrophils | Day 30
  Neutrophil concentration in peripheral blood (cells/µL)
Peripheral blood flow cytometry - neutrophils | Day 300
  Neutrophil concentration in peripheral blood (cells/µL)
Survival | baseline to 24 months
  Survival and time to death/cause of death (if applicable) of study subjects

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan A Galli, MD, Principal Investigator — Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thabut G, Mal H, Castier Y, Groussard O, Brugiere O, Marrash-Chahla R, Leseche G, Fournier M. Survival benefit of lung transplantation for patients with idiopathic pulmonary fibrosis. J Thorac Cardiovasc Surg. 2003 Aug;126(2):469-75. doi: 10.1016/s0022-5223(03)00600-7. PMID 12928646
- [Background] Lund LH, Edwards LB, Dipchand AI, Goldfarb S, Kucheryavaya AY, Levvey BJ, Meiser B, Rossano JW, Yusen RD, Stehlik J; International Society for Heart and Lung Transplantation. The Registry of the International Society for Heart and Lung Transplantation: Thirty-third Adult Heart Transplantation Report-2016; Focus Theme: Primary Diagnostic Indications for Transplant. J Heart Lung Transplant. 2016 Oct;35(10):1158-1169. doi: 10.1016/j.healun.2016.08.017. Epub 2016 Aug 21. No abstract available. PMID 27772668
- [Background] Schaffer JM, Singh SK, Reitz BA, Zamanian RT, Mallidi HR. Single- vs double-lung transplantation in patients with chronic obstructive pulmonary disease and idiopathic pulmonary fibrosis since the implementation of lung allocation based on medical need. JAMA. 2015 Mar 3;313(9):936-48. doi: 10.1001/jama.2015.1175. PMID 25734735
- [Background] Elicker BM, Golden JA, Ordovas KG, Leard L, Golden TR, Hays SR. Progression of native lung fibrosis in lung transplant recipients with idiopathic pulmonary fibrosis. Respir Med. 2010 Mar;104(3):426-33. doi: 10.1016/j.rmed.2009.10.019. Epub 2009 Nov 12. PMID 19913395
- [Background] Wahidi MM, Ravenel J, Palmer SM, McAdams HP. Progression of idiopathic pulmonary fibrosis in native lungs after single lung transplantation. Chest. 2002 Jun;121(6):2072-6. doi: 10.1378/chest.121.6.2072. PMID 12065382
- [Background] Wollin L, Wex E, Pautsch A, Schnapp G, Hostettler KE, Stowasser S, Kolb M. Mode of action of nintedanib in the treatment of idiopathic pulmonary fibrosis. Eur Respir J. 2015 May;45(5):1434-45. doi: 10.1183/09031936.00174914. Epub 2015 Mar 5. PMID 25745043
- [Background] Xu Z, Ramachandran S, Gunasekaran M, Zhou F, Trulock E, Kreisel D, Hachem R, Mohanakumar T. MicroRNA-144 dysregulates the transforming growth factor-beta signaling cascade and contributes to the development of bronchiolitis obliterans syndrome after human lung transplantation. J Heart Lung Transplant. 2015 Sep;34(9):1154-62. doi: 10.1016/j.healun.2015.03.021. Epub 2015 Mar 27. PMID 25979625
- [Background] Sjoland AA, Callerfelt AK, Thiman L, et al. Prostacyclin and VEGF in the rejection process after lung transplantation-A possible biomarker [abstract]. Eur Respir J. 2016; PA4040.
- [Background] Suhling H, Bollmann B, Gottlieb J. Nintedanib in restrictive chronic lung allograft dysfunction after lung transplantation. J Heart Lung Transplant. 2016 Jul;35(7):939-40. doi: 10.1016/j.healun.2016.01.1220. Epub 2016 Feb 9. No abstract available. PMID 26996931
- [Background] Delanote I, Wuyts WA, Yserbyt J, Verbeken EK, Verleden GM, Vos R. Safety and efficacy of bridging to lung transplantation with antifibrotic drugs in idiopathic pulmonary fibrosis: a case series. BMC Pulm Med. 2016 Nov 18;16(1):156. doi: 10.1186/s12890-016-0308-z. PMID 27863518
- [Background] Dorey-Stein Z, Galli JA, Criner GJ. Effect of antifibrotic therapy in patients with idiopathic pulmonary fibrosis awaiting lung transplantation [abstract]. Am J Respir Crit Care Med. 2017;195:A5386
- [Background] Leuschner G, Stocker F, Veit T, Kneidinger N, Winter H, Schramm R, Weig T, Matthes S, Ceelen F, Arnold P, Munker D, Klenner F, Hatz R, Frankenberger M, Behr J, Neurohr C. Outcome of lung transplantation in idiopathic pulmonary fibrosis with previous anti-fibrotic therapy. J Heart Lung Transplant. 2017 Jul 5:S1053-2498(17)31886-7. doi: 10.1016/j.healun.2017.07.002. Online ahead of print. PMID 28734935